CLINICAL TRIAL: NCT05614713
Title: Effect of Sensory Integration Therapy on Balance and Functional Mobility in Children With Spastic Cerebral Palsy
Brief Title: Effect of Sensory Integration Therapy on Balance and Functional Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elsayed Abbass, Mai Elsayed Abbass, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003289
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: study group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): received a modified selected physical therapy program to increase sensory input.
  Interventions: Procedure: Modified physical therapy program to increase sensory input
- Control group (Active Comparator): received a selected physical therapy
  Interventions: Procedure: Selected physical therapy program

INTERVENTIONS:
Procedure: Selected physical therapy program — Gait training and balance training
  Arms: Control group
Procedure: Modified physical therapy program to increase sensory input — Gait training and balance training using sensory stimulating matts
  Arms: Study group

SUMMARY:
Purpose: to investigate the effect of sensory integration therapy on balance and functional mobility in children with spastic diplegic cerebral palsy. Methods: children with spastic cerebral palsy, the children were assigned to a control group and a study group. Balance was assessed using the Biodex balance system and functional mobility was assessed using the Timed Up and Go test.

DETAILED DESCRIPTION:
Purpose: to investigate the effect of sensory integration therapy on balance and functional mobility in children with spastic diplegic cerebral palsy. Methods: children with spastic cerebral palsy, the children were assigned to a control group and a study group. Balance was assessed using the Biodex balance system and functional mobility was assessed using the Timed Up and Go test. The control group received selected physical therapy, while the study group received the previously mentioned selected physical therapy program modified to increase sensory input. Treatment sessions for both groups were conducted for both groups for 1 hour once a day, three times per week for two successive months.

ELIGIBILITY:
Inclusion Criteria:

Ages from 6-10 years old. The degree of spasticity was 1 to 1+ Level II according to the Gross motor function classification system

Exclusion Criteria:

Visual or auditory problems. Fixed deformities of lower limbs.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Assessment of balance | After 2 months of intervention
  Assessment by using Biodex Balance System
Assessment of functional mobility | After 2 months of intervention
  Assessment by using the Timed Up and Go test

CONTACTS AND LOCATIONS:
Overall Officials: Mai E Abbass, Ph.D., Study Director — Cairo University
Locations (1):
- Faculty of physical therapy, Cairo university, Cairo, Egypt